CLINICAL TRIAL: NCT07095179
Title: Acute Effects of Intermittent Inspiratory Muscle Training on Blood Glucose and Vascular Function Responses
Brief Title: Effects of Inspiratory Muscle Exercise on Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202506HM022
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Intermittent Inspiratory Muscle Training; Eupnea
Keywords: Energy Expenditure; Metabolic Health; Pulse Wave Velocity; Inspiratory muscle training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eupnea (Experimental): Participants will breathe normally.
  Interventions: Behavioral: Eupnea
- Inspiratory muscle training (Experimental): Intermittent inspiratory muscle training (IMT) will be conducted throughout the trial
  Interventions: Behavioral: Intermittent inspiratory muscle training (IIMT)

INTERVENTIONS:
Behavioral: Eupnea — Participants will breathe normally.
  Arms: Eupnea
Behavioral: Intermittent inspiratory muscle training (IIMT) — Intermittent inspiratory muscle training (IIMT) will be conducted throughout the trial
  Arms: Inspiratory muscle training

SUMMARY:
The purpose of this study is to investigate whether inspiratory muscle training has an immediate effect on energy expenditure, heart rate, blood glucose, blood pressure, and arterial stiffness in healthy adults, obese adults, and adults with type 2 diabetes.

DETAILED DESCRIPTION:
Participants will be asked to complete two trials involving intermittent exercise, which will include eupnea and inspiratory muscle training (IMT), as well as a resting control condition, in a randomized crossover study design. The trials will be separated by a minimum of 48 hours and will be completed within a 7-day period. Throughout all trials, participants will be required to remain relaxed and seated on an adjustable examination bed. For the IMT intensity, participants will utilize an inspiratory muscle training device (PowerBreathe Plus, Powerbreathe International Ltd., UK) and adjust the resistance to a level at which breathing continuously for 20 breaths is perceived as "somewhat hard" (RPE = 13), according to the Rating of Perceived Exertion (RPE) scale. This will take place during a 3.5-hour oral glucose tolerance test (OGTT). During the trials, participants may watch television or read; however, typing on a laptop or computer will be prohibited.

ELIGIBILITY:
Inclusion Criteria

* Healthy adults, obese adults and adults with type 2 diabetes
* Aged between 20 to 45 years
* Weight stable for more than 3 months (no change in weight +/- 3%)
* Non-smoker
* Non-highly trained athletic team members
* Normal lifestyle patterns

Exclusion Criteria

* Personal history of/existing hypertension, respiratory infectious disease, cardiovascular disease, metabolic disease
* Taking medications that may influence lipid or carbohydrate metabolism or immune system function

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood glycaemic responses | 0 (baseline), 30, 60, 120, and 210 minutes during the 210-minute trial
  Changes in blood glycaemic responses between trials
Pulse wave velocity (PWV) | 0 (baseline), 30, 60, 90, 150, and 210 minutes during the 210-minute trial
  Changes in pulse wave velocity between trials

SECONDARY OUTCOMES:
Energy expenditure | First 90 minutes during the 210-minute trial
  Changes in energy expenditure between trials
Heart Rate Variability (HRV) | In a regular patterns during the 210-minute trial
  Changes in Heart Rate Variability (HRV) between trials
Visual analogue scale (VAS) | Every 30 minutes during the 210-minute trial
  Changes in the visual analogue scale (VAS) ranged from 0 to 100 mm, with higher values indicating a greater intensity of sensation between trials.
Perceived stress scale (PSS) | Every 30 minutes during the 210-minute trial
  Changes in perceived stress scale (PSS) with higher values indicating a greater intensity of sensation between trials.